CLINICAL TRIAL: NCT03730857
Title: Early Predictors of Poor Treatment Response in Patients With Schizophrenia Treated With Atypical Antipsychotics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calo Psychiatric Center (Other)
Responsible Party: Principal Investigator, For-Wey Lung, Superintendent and Attending physician, Calo Psychiatric Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: T1-02
Record Dates: First submitted 2018-10-31; First posted 2018-11-05 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; PANSS; positive predictive value; negative predictive value
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine; Risperidone; Paliperidone Palmitate

STUDY DESIGN:
Intervention Model Description: One hundred eleven inpatients with acutely exacerbated schizophrenia were randomized to give optimal therapy of olanzapine, risperidone, and paliperidone in one-week run-in period and 12 weeks' intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- olanzapine (Active Comparator): olanzapine has a dose of 10 to 20 mg daily for 12 weeks
  Interventions: Drug: Olanzapine
- risperidone (Active Comparator): risperidone at a dose of 4 to 6 mg daily for 12 weeks
  Interventions: Drug: risperidone
- paliperidone (Active Comparator): paliperidone at a dose of 6 to 12 mg daily for 12 weeks.
  Interventions: Drug: Paliperidone

INTERVENTIONS:
Drug: Olanzapine — olanzapine tablet
  Other Names: second-generation antipsychotics
  Arms: olanzapine
Drug: risperidone — risperidone tablet
  Other Names: second-generation antipsychotics
  Arms: risperidone
Drug: Paliperidone — paliperidone tablet
  Other Names: second-generationantipsychotics
  Arms: paliperidone

SUMMARY:
Background: The aims of this study were to explore the relationship between early reduction in psychotic symptoms and the ultimate response in patients with schizophrenia treated by atypical antipsychotics, and to determine the best time to switch or maitain the regimen. PI also explore the possible predictors for the clinical response.

Methods: One hundred eleven inpatients with acutely exacerbated schizophrenia were randomized to give optimal therapy of olanzapine, risperidone, and paliperidone in one-week run-in period and 12 weeks' intervention. All participants were assessed using Positive and Negative Syndrome Scale (PANSS). Early Response, defined as reduction of 25% in PANSS score, was examined at weeks 1, 2, 3, 4 and 8, and these ratings were used to predict ultimate response (25% PANSS reduction) at week 12. PI hypothesized that early treatment response at Week 1 or 2 could predict Week 12's treatment outcome.

DETAILED DESCRIPTION:
Study Design: This study recruited hospitalized adult patients who had a relapse of schizophrenia. All participants had received antipsychotic treatment for a period of time previously. They have to meet the diagnostic criteria for schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV). One hundred and twenty adult inpatients were recruited and were randomly assigned to receive olanzapine (n=60), risperidone (n=30) and paliperidone (n=30) in an allocation ratio of 2:1:1. The participants were allowed to change the dosage of antipsychotics and their hospitalization status according to the judgement of in-charged physicians during the study period.

The study was approved by the Institutional Review Board and written informed consents were obtained either directly from the patients or from their legal guardians after the study had been explained. The inclusion criteria for this study were: (1) age 18 to 65 years, (2) no major systemic illnesses based on physical examinations and laboratory test results, and (3) baseline PANSS total score≧60. The exclusion criteria were as follows: (1) participants not taking any antipsychotics in the previous one month, (2) participants were pregnant and lactating women, and (3) history of clozapine treatment in the previous 3 months, and (4) patients receiving long-acting antipsychotic injections in the preceding 6 months of enrollment.

This study was conducted by a 12-week, open-label and naturalistic randomized design. A tri-therapy (olanzapine, risperidone, and paliperidone) completely randomized design was adopted for this study, which involved three homogeneous groups of patients with a run-in period of 3 months. The patients were required to have discontinued all prior use of antipsychotics for a period of at least 7 days before their entry into the study. During wash-out period, administration of either oral benzodiazpines, hypnotics or injection of lorazepam to control anxiety, insomnia and aggression were allowed. After the wash-out period, the patients received treatment with an atypical antipsychotic drug, olanzapine, risperidone or paliperidone for 3 months.

The Positive and Negative Syndrome Scale (PANSS) rating scale was used to evaluate the changes of psychiatric symptoms in each time point. The subject patients were interviewed for the PANSS by senior psychiatrists. The raters in the present study had worked mainly on inpatient treatment of severe schizophrenic patients, and were well acquainted with symptoms of schizophrenia. Prior to the present study, all participating psychiatrists had received adequate training through the manual and they had had clinical experience in the PANSS rating before the study. At each time point if the scores of PANSS showed the patient's symptoms had worsened, the dosage would be adjusted based on the clinical judgment of in-charged senior psychiatrist. However, if the scores of PANSS were improved, the dosage was maintained. The recommended dose for the three groups were as follows: 10 to 20 mg daily for olanzapine, 4 to 6 mg daily for risperidone, and 6 to 12 mg daily for paliperidone. Throughout the study period, the paticipants were allowed to continuously use some concomitant medication, including lorazepam (up to 6 mg/day) for insomnia or agitation and biperiden (up to 6 mg/day) for treatment of extrapyramidal side effects. No other psychotropic agents were administered during the 12-week study.

ELIGIBILITY:
Inclusion Criteria:

* (1) age 18 to 65 years,
* (2) no major systemic illnesses based on physical examinations and laboratory test results,
* (3) baseline PANSS total score≧60

Exclusion Criteria:

* (1) participants not taking any antipsychotics in the previous one month,
* (2) participants were pregnant and lactating women,
* (3) history of clozapine treatment in the previous 3 months,
* (4) patients receiving long-acting antipsychotic injections in the preceding 6 months of enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 12 weeks
  The Positive and Negative Syndrome Scale (PANSS) rating scale was used to evaluate the changes of psychiatric symptoms in each time point. The raters in the present study had worked mainly on inpatient treatment of severe schizophrenic patients, and were well acquainted with symptoms of schizophrenia.

CONTACTS AND LOCATIONS:
Overall Officials: For-Wey Lung, MD, ScD, Principal Investigator — Calo Psychiatric Center

REFERENCES:
- [Derived] Chen YL, Chen KP, Chiu CC, Tai MH, Lung FW. Early predictors of poor treatment response in patients with schizophrenia treated with atypical antipsychotics. BMC Psychiatry. 2018 Dec 4;18(1):376. doi: 10.1186/s12888-018-1950-1. PMID 30509308